CLINICAL TRIAL: NCT05487924
Title: Stroke Volume Variation- Guided Hemodynamic Therapy Versus Oxygen Extraction Ratio-guided Hemodynamic Therapy on Outcomes Following Laparoscopic Gastrointestinal Cancer Surgery
Brief Title: Stroke Volume Variation- Guided Hemodynamic Therapy Versus Oxygen Extraction Ratio-guided Hemodynamic Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, YANXIA SUN, Principal Investigator, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BJH-005
Record Dates: First submitted 2022-07-24; First posted 2022-08-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Goal-directed Fluid Therapy
Keywords: stroke volume variation; oxygen extraction ratio; goal-directed fluid therapy; laparoscopic gastrointestinal surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SVV-GDHT (Experimental): SVV ≤12% and CI of at least 2.5 L•min-1•m-2 were required. 500 mL of crystalloids was infused during induction, followed by a 2 ml•kg-1•h-1continuous infusion. If SVV was higher than 12% for over 5 minutes, a 250 mL bolus of crystalloid was given. Another 250 ml bolus of colloid was administrated if SVV was still higher than 12% or SVV decreased over 10%. If CI value was below 2.5 L•min-1•m-2, inotropes were applied to reach this minimum CI, serving as a safety parameter to prevent patients from low cardiac output. If SVV and CI were within the target range but MAP was below 65 mmHg, norepinephrine was started. After the initial assessment, patients were reassessed every 5 minutes intraoperatively to maintain values according to the study algorithm
  Interventions: Other: SVV-GDHT
- O2ER-GDHT (Experimental): the goal of O2ER is assessed every one hour to keep O2ER<27% which calculated by the following equation:(SaO2 - SvO2)/SaO2, when O2ER is greated than 27%, CVP lower than 10mmHg, 250ml colloid is given, otherwise, inotropes is given as CVP≥10mmHg.
  Interventions: Other: O2ER-GDHT
- conventional care (Active Comparator): MAP was kept between 65 and 90 mmHg, CVP between 8 and 12 mmHg and urinary output more than 0.5 ml•kg-1•h-1. 500 ml of crystalloids was infused during induction, followed by a continuous infusion of crystalloids (4 ml•kg-1•h-1). If the MAP decreased below 65 mmHg, or if the CVP decreased below 8 mmHg, a 250 mL bolus of colloid was given after waiting 5 minutes if any one of the criteria was met. If the MAP decreased below 65 mmHg and remained unresponsive to fluids, norepinephrine or inotropes was given to maintain the MAP above 65 mmHg.
  Interventions: Other: conventional care

INTERVENTIONS:
Other: SVV-GDHT — GDHT guided by SVV using Flotra/Vigileo monitor
  Arms: SVV-GDHT
Other: O2ER-GDHT — GDHT guided by O2ER
  Arms: O2ER-GDHT
Other: conventional care — conventional fluid therapy without GDHT
  Arms: conventional care

SUMMARY:
The FloTrac/Vigileo is a minimal invasive device assessing flow based hemodynamic parameters by pulse contour analysis based on the radial artery pressure signal. This method gained popularity as it is minimally invasive compared to esophageal Doppler or pulmonary artery catheter insertion and provides continuous beat-to-beat data. The previous study with 110 patients found that that GDHT guided by stroke volume variation (SVV) using the FloTrac/Vigileo device was associated with a reduced length of hospital stay and a lower incidence of POGD in major abdominal oncological surgery. However, no difference was found in the incidence of postoperative complications between the two groups, lack of statistical power could be a limitation to demonstrate the true association. Therefore, further prospective trials are needed to address this issue.

The use of early and efficient therapeutic strategies able to detect and to treat potential triggers of organ failures, such as tissue hypoperfusion, is particularly important. If hypoperfusion is not adequately managed, tissue hypoxia could occur, resulting from an impairment of the adaptive mechanisms of myocardial contractile function, under the influence of inflammatory mediators, and the peripheral tissues will then increase their oxygen extraction (O2ER). AS such, GDHT guided by O2ER may be appropriate to monitor GDHT strategies because it reflects the balance between oxygen delivery and consumption.

Therefore, the investigators performed this single-center, randomized, controlled trial to investigate whether GDHT guided by SVV using FloTrac/Vigileo monitor and GDHT guided by O2ER would reduce incidence of postoperative complication and shorten the length of hospital stay, compared with a standard conventional fluid therapy in low-to-moderate risk patients undergoing major laparoscopic gastrointestinal oncological surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18~80 years
2. ASA I~III
3. Patients undergoing elective major laparoscopic gastrointestinal oncological surgery.Procedures were considered major if listed for resection cancer with tumor debulking, staging or reconstruction with a risk for significant surgical blood loss.

Exclusion Criteria:

1. co-existing congestive heart failure; chronic lung disease; or renal or hepatic dysfunction (creatinine >50 % or liver enzymes >50 % of normal values), and arrhythmias.
2. less than 18 years
3. pregnant or lactating woman
4. patients undergoing emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative complication | 30 days after surgery
  the number of patients with predefined moderate or major postoperative complications (pulmonary embolism, myocardial ischemia or infarction, arrhythmia, cardiac or respiratory arrest, limb or digital ischemia, cardiogenic pulmonary edema, acute respiratory distress syndrome, gastrointestinal bleeding, bowel infarction, anastomotic breakdown, paralytic ileus, acute psychosis, stroke, acute kidney injury, infection [source uncertain], urinary tract infection, surgical site infection, organ/space infection, bloodstream infection, nosocomial pneumonia, and postoperative hemorrhage

SECONDARY OUTCOMES:
Length of hospital stay | from the end of surgery until the date of discharge from hospital,assessed up to 30 days after surgery
  Length of stay was determined by the period from completion of surgery to discharge
critical care-freedays | 30 days after surgery
  numberof days alive and not in critical care
mortality | all-cause mortality at 30 days following surgery; all-cause mortality at 180 days following surgery
  all cause mortality
postoperative recovery quality | 1, 3, 7 days after surgery
  QoR15, 0 :not at all , 10: most of time
time to first tolerate of an oral diet | from the end of surgery until the date of discharge from hospital,assessed up to 30 days after surgery
  time from the end of surgery and first tolerate of an oral diet
time to first flatus | from the end of surgery until the date of discharge from hospital,assessed up to 30 days after surgery
  duration between the end of surgery and first flatus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol